CLINICAL TRIAL: NCT03416504
Title: A Translational Study of the Mechanisms of Exposure Therapy for Obsessions: Gradual vs. Variable Exposure Intensity
Brief Title: Methods for Managing Intrusive Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Association for Behavioral and Cognitive Therapies (ABCT) (Unknown); American Psychological Association (APA) (Other)
Responsible Party: Principal Investigator, Jon Abramowitz, PhD, Professor, Clinical Psychology, Department of Psychology and Neuroscience, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-3310; 5101599 (Other: ABCT); 5103050 (Other: APA)
Record Dates: First submitted 2018-01-21; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either gradual or variable exposure
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators were blind to the exposure condition participants were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gradual Exposure Group (Experimental): The gradual exposure group received the Gradual Exposure (EXP-G) Intervention.
  Interventions: Behavioral: Gradual Exposure (EXP-G)
- Variable Exposure Group (Experimental): The variable exposure group received the Variable Exposure (EXP-V) Intervention.
  Interventions: Behavioral: Variable Exposure (EXP-V)

INTERVENTIONS:
Behavioral: Gradual Exposure (EXP-G) — In EXP-G, exposure proceeded hierarchically from mildly, to moderately, to highly intense stimuli so that exposure intensity gradually built between (but not within) sessions.
  Arms: Gradual Exposure Group
Behavioral: Variable Exposure (EXP-V) — In EXP-V, exposure stimuli were chosen at random (i.e., pieces of paper with exposure stimuli written on them were pulled randomly from an opaque container) so that mild, moderate, and high intensity exposures could occur in any order during any of the sessions (the participant was not informed which level was coming next). This aimed to maximize (a) uncertainty, (b) variability in exposure intensity, and (c) variability in corresponding physiological arousal.
  Arms: Variable Exposure Group

SUMMARY:
The current study sought to translate laboratory research on learning and memory to better understand the mechanisms and methods for implementing exposure therapy for unwanted obsessional thoughts. Specifically, we compared the processes and the short- and long-term outcomes of: (a) gradual exposure (EXP-G), emphasizing hierarchical exposure completion, versus (b) variable exposure (EXP-V), emphasizing variability in exposure intensity.

DETAILED DESCRIPTION:
Although preliminary research suggests that learning to tolerate varying levels of fear during exposure enhances outcomes for some anxiety-related problems, no previous study has examined this possibility in the context of unwanted obsessions. Adults with a moderately distressing obsessional thought were randomly assigned to four twice-weekly sessions of either: (a) gradual exposure (EXP-G), emphasizing hierarchical exposure completion, or (b) variable exposure (EXP-V), emphasizing variability in exposure intensity.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Willing to attend and audiotape all study sessions
* Fluent in English
* Presence of one or more obsessional thoughts that cause marked distress
* If on a psychiatric medication (e.g., SSRI), willing to remain at a fixed dose while participating in the study (and stabilized on medication for 30 days before beginning the intervention).

Exclusion Criteria:

* Previous cognitive behavioral therapy (CBT) for anxiety
* Current suicidal ideation
* Current substance use disorder
* Current mania or psychosis
* Currently taking an anxiolytic (e.g., Ativan) or stimulant (e.g., Ritalin) medication
* Heart, respiratory, or neurological condition
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score at 3-month follow-up (week 14) | Baseline (week 0) and 3-month follow-up (week 14)
  The Y-BOCS is a clinician-administered interview that assesses obsessive compulsive disorder (OCD) symptom severity over the past week. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).

SECONDARY OUTCOMES:
Change from baseline in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score at post-treatment (week 2) | Baseline (week 0) and post-treatment (week 2)
  The Y-BOCS is a clinician-administered interview that assesses obsessive compulsive disorder (OCD) symptom severity over the past week. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).
Changes from baseline in Dimensional Obsessive-Compulsive Scale-Unacceptable Thoughts (DOCS-UT) at 3-month follow-up (week 14) | Baseline (week 0) and 3-month follow-up (week 14)
  The DOCS-UT is a self-report measure of the clinical severity of the unwanted thoughts (UT) OCD symptom dimension. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).
Changes from baseline in Dimensional Obsessive-Compulsive Scale-Unacceptable Thoughts (DOCS-UT) at post-treatment (week 2) | Baseline (week 0) and post-treatment (week 2)
  The DOCS-UT is a self-report measure of the clinical severity of the unwanted thoughts (UT) OCD symptom dimension. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).
Changes from baseline in Behavioral Approach Test (BAT) Mean Subjective Units of Distress (SUDS) at 3-month follow-up (week 14) | Baseline (week 0) and 3-month follow-up (week 14)
  The BAT is an in vivo measure of participants' behavioral responses to their target obsession. Participant SUDS were collected for 5 increasingly difficult steps participants completed related to their obsessional thought. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).
Changes from baseline in Behavioral Approach Test (BAT) Mean Subjective Units of Distress (SUDS) at post-treatment (week 2) | Baseline (week 0) and post-treatment (week 2)
  The BAT is an in vivo measure of participants' behavioral responses to their target obsession. Participant SUDS were collected for 5 increasingly difficult steps participants completed related to their obsessional thought. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).
Changes from baseline in Behavioral Approach Test (BAT) Number of Steps Completed at 3-month follow-up (week 14) | Baseline (week 0) and 3-month follow-up (week 14)
  The BAT is an in vivo measure of participants' responses to their target obsession. The number of steps participants were able to complete without performing a ritual were calculated. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).
Changes from baseline in Behavioral Approach Test (BAT) Number of Steps Completed at post-treatment (week 2) | Baseline (week 0) and post-treatment (week 2)
  The BAT is an in vivo measure of participants' responses to their target obsession. The number of steps participants were able to complete without performing a ritual were calculated. This measure will be used to assess change over the course of the intervention at four time-points throughout the study (over approximately 3.5 months total).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Abramowitz, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacoby RJ, Abramowitz JS, Blakey SM, Reuman L. Is the hierarchy necessary? Gradual versus variable exposure intensity in the treatment of unacceptable obsessional thoughts. J Behav Ther Exp Psychiatry. 2019 Sep;64:54-63. doi: 10.1016/j.jbtep.2019.02.008. Epub 2019 Feb 26. PMID 30851653